CLINICAL TRIAL: NCT00127582
Title: Evaluation of Arrhythmic Risk in Myotonic Dystrophy Type I (DM 1)
Brief Title: RAMYD Study - Evaluation of Arrhythmic Risk in Myotonic Dystrophy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione Telethon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUP02067
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Last update posted 2005-08-25 (Estimated); Status verified 2005-05

CONDITIONS: Myotonic Dystrophy; Sudden Cardiac Death
Keywords: Myotonic dystrophy type 1; Sudden cardiac death; Ventricular tachyarrhythmias; Bradyarrhythmias
MeSH Terms: conditions — Myotonic Dystrophy; Death, Sudden, Cardiac; Tachycardia, Ventricular; Bradycardia | interventions — Mutagenesis, Insertional; Defibrillators, Implantable

INTERVENTIONS:
Procedure: Electrophysiological study
Device: pacemaker (PM) implant, internal cardiac defibrillator (ICD) implant, loop-recorder implant

SUMMARY:
This is a prospective multicentric Italian study to evaluate the arrhythmic risk in myotonic dystrophy type 1.

DETAILED DESCRIPTION:
Myotonic dystrophy type 1 (DM1, Steinert disease) is a multisystem disorder that affects, beside muscle, several other organs, including the heart.

Cardiac involvement represents a major problem in the clinical management of patients, so that cardiac complications represent one of the primary causes of premature death in DM1. In particular there is a high incidence of sudden death, ranging from 2 to 30% of cases, so far principally related to the development of conduction blocks. However, literature reports of sudden death in patients implanted with pacemakers, as well as of spontaneous ventricular tachycardia would suggest a potential etiologic role also for ventricular arrhythmias. The lack of clinical research studies conducted on a large number of patients does not make available definite data regarding the etiology and the epidemiology of arrhythmic events in DM1. For the same reasons, other considerable topics, such as prognostic stratification of the arrhythmic risk and clinical management of life-threatening arrhythmias in DM1 patients, are still undefined.

To clarify these issues, the investigators propose a clinical research study performed on a large cohort of DM1 patients enrolled through a multicenter collaboration that also involves 5 cardiological-neurological Italian centres.

Aims of this study are:

* To estimate the incidence of arrhythmias and to characterize the brady-tachyarrhythmic mechanisms underlying the occurrence of cardiac sudden death in DM1;
* To verify by statistical analysis the reliability of data obtained from both non invasive and invasive diagnostic procedures as indexes useful for estimating the arrhythmic risk in DM1;
* To identify more adequate therapeutic guidelines in order to prevent the occurrence of life-threatening arrhythmias.

The protocol of study includes:

1. Clinical-genetic evaluation;
2. Non invasive and invasive diagnostic cardiac procedures;
3. The use of devices for diagnostic and therapeutic follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected by myotonic dystrophy type I (MD1).
* Patient willing to provide a signed informed consent.

Exclusion Criteria:

* Age < 18 years old or >70 years old.
* Ischemic cardiomyopathy
* Cardiomyopathy due to chronic excess of alcohol consumption (>100 g\day)
* Congenital heart disease
* Acquired valvular heart disease
* Metabolic cardiomyopathy: thyrotoxicosis, hypothyroidism, adrenal cortical insufficiency, pheochromocytoma, acromegaly
* Familiar storage and infiltrative diseases (hemochromatosis, glycogen storage, Hurler's syndrome, Niemann-Pick disease; primary, secondary, familial and hereditary cardiac amyloidoses)
* Systemic diseases (connective tissue disorder; sarcoidosis)
* Peripartum cardiomyopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537
Dates: Start 2003-01

PRIMARY OUTCOMES:
Evaluate incidence of: major cardiac events (sudden death
resuscitated cardiac arrest
ventricular fibrillation
sustained ventricular tachycardia
sinoatrial and atrioventricular [AV] blocks)

SECONDARY OUTCOMES:
Evaluate with diagnostic non-invasive (standard electrocardiogram [ECG]
24-hour monitoring ECG
signal-averaged ECG
echocardiography) and invasive procedures (electrophysiology study [EPS] and implantable loop recorders) the risk to develop cardiac arrhythmias in DM patients

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Bellocci, MD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Rome, Italy

REFERENCES:
- [Background] Pelargonio G, Dello Russo A, Sanna T, De Martino G, Bellocci F. Myotonic dystrophy and the heart. Heart. 2002 Dec;88(6):665-70. doi: 10.1136/heart.88.6.665. No abstract available. PMID 12433913
- [Derived] Dello Russo A, Mangiola F, Della Bella P, Nigro G, Melacini P, Bongiorni MG, Tondo C, Calo L, Messano L, Pace M, Pelargonio G, Casella M, Sanna T, Silvestri G, Modoni A, Zachara E, Moltrasio M, Morandi L, Nigro G, Politano L, Palladino A, Bellocci F. Risk of arrhythmias in myotonic dystrophy: trial design of the RAMYD study. J Cardiovasc Med (Hagerstown). 2009 Jan;10(1):51-8. doi: 10.2459/jcm.0b013e328319bd2c. PMID 19708226